CLINICAL TRIAL: NCT00380341
Title: Effects of Instrument-Applied Spinal Manipulative Therapy on Postureal Control and Autonomic Balance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Logan College of Chiropractic (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RD0803050033
Record Dates: First submitted 2006-09-21; First posted 2006-09-25 (Estimated); Last update posted 2008-10-17 (Estimated); Status verified 2008-10

CONDITIONS: Heart Rate

INTERVENTIONS:
Procedure: Instrument-applied spinal manipulative therapy

SUMMARY:
The purpose of this study is to determine the effects of spinal manipulative therapy on autonomic balance and to determine if there exists a relationship between autonomic state and postural control.

DETAILED DESCRIPTION:
Previous studies have demonstrated that sensory and cognitive systems share some common neural substrate. The afferent neural impuleses of mechanoreception (also known as somatosensation) as produced by joint mechanoreceptors and adjacent muscle spindle cells may impact supraspinal centers. Few studies have been done to determine if the afferent impulses generated by spinal manipulative therapy (SMT) can impact the porcessing that occurs at supra-spinal centers. The relationship between postural control and cognition is studies using a dual-tak methodology, a primary (postural) task will often demonstrate degradation with the addition of a secondary, concurrent (cognitive) task. The current study seeks to determine the effects of SMT on postrual control using a dual-task paradigm, while monitoring autonomic state (using Heart Rate Variability analysis) during the course of therapy. It is thought that SMT can improve HRV status, and postural control within a dual-task situation, and that there will be differences in postural control related to a participant's HRV status. Activities of daily living often invole the coupling of a cognitive task with a complex postural task.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults currently enrolled at Logan College

Exclusion Criteria:

* Lower extremity injury, vestibular disorders

Ages: 19 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20
Dates: Start 2006-09; Study Completion 2006-11

CONTACTS AND LOCATIONS:
Overall Officials: Kristan J. Giggey, DC, Principal Investigator — Logan College of Chiropractic; Rodger Tepe, PhD, Study Director — Logan College of Chiropractic